CLINICAL TRIAL: NCT03720756
Title: Effect of a Nickel Free Diet and Nickel Sensitization on GERD Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Zachary Zinn, Program Director, Assistant Professor of Dermatology, West Virginia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1804080531
Record Dates: First submitted 2018-10-05; First posted 2018-10-25 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Gastroesophageal Reflux
Keywords: nickel-free; diet; GERD; Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Patients will undergo a patch test to determine if they are hypersensitive to nickel among other metabolites. Regardless of the results of the patch test, patients will be placed on a nickel-free diet for 8 weeks.
Who Masked: Participant
Masking Description: The efficacy of treatment methods will be assessed by comparing GERD-Health Related Quality of Life (HRQL) questionnaires before and after implementation of a nickel-free diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects WITH nickel-sensitivity (Experimental): Subjects on nickel-free diet who have a positive patch-test result, indicating nickel-sensitivity.
  Interventions: Other: Nickel-free diet
- Subjects WITHOUT nickel-sensitivity (Active Comparator): Subjects on nickel-free diet who have a negative patch-test result, indicating they do NOT have nickel-sensitivity.
  Interventions: Other: Nickel-free diet

INTERVENTIONS:
Other: Nickel-free diet — Subjects follow a nickel-free diet. Lists of acceptable foods will be provided to subjects.

SUMMARY:
There is little evidence on the effect of a nickel-free diet on gastroesophageal reflux disease (GERD). We hope to determine if a nickel-free diet improves GERD symptoms in patients with a nickel allergy by having patients complete a questionnaire on their GERD symptoms before and after initiation of 8 weeks on a nickel-free diet.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older with a history of GERD
* owns a phone with a camera
* has access to or is willing to sign up for MyChart
* is symptomatic for GERD at time of visit as determined by a score of >12 on the GERD Health Related Quality of Life (GERD-HRQL) questionnaire. (Patients that are currently taking a proton pump inhibitor (PPI) they must have been on the PPI for at least 3 months.)

Exclusion Criteria:

* less than 18 years of age
* no not have access to MyChart
* are not willing to sign up for MyChart
* have taken an oral steroid within 4 weeks
* have experienced a sunburn or had significant sun exposure within the last 4 weeks, or applied a topical steroid to the area that the past test will be applied (i.e. upper back or arm) in the last 4 weeks. No vulnerable populations will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Change in baseline Gastroesophageal reflux disease-Health Related Quality of Life (GERD-HRQL) Questionnaire score | after 8 weeks on nickel-free diet
  questionnaire to assess severity of GERD. Total Score: Calculated by summing the individual scores to questions 1-12. Greatest possible score (worst symptoms) = 60; Lowest possible score (no symptoms) = 0. For the purposes of our study, a score of 13 or above is considered symptomatic for GERD.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - WVU Medicine University Town Center, Morgantown, West Virginia
  - Physician's Office Center at Ruby Memorial, Digestive Diseases, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No
We do not plan to make IPD available to other researchers.

REFERENCES:
- [Derived] Yousaf A, Hagen R, Mitchell M, Ghareeb E, Fang W, Correa R, Zinn Z, Gayam S. The effect of a low-nickel diet and nickel sensitization on gastroesophageal reflux disease: A pilot study. Indian J Gastroenterol. 2021 Apr;40(2):137-143. doi: 10.1007/s12664-020-01090-3. Epub 2020 Nov 21. PMID 33219986